CLINICAL TRIAL: NCT01919801
Title: Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Clinical Study Evaluating the Safety & Efficacy of Icatibant as a Treatment for Angiotensin-Converting Enzyme Inhibitor (ACE-I)-Induced Angioedema in Adults
Brief Title: Blinded Safety & Efficacy Placebo Controlled Study of Icatibant for Angiotensin Converting Enzyme Inhibitor Induced Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGT-FIR-096; 2014-001213-12 (EudraCT Number)
Record Dates: First submitted 2013-07-25; First posted 2013-08-09 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Angiotensin Converting Enzyme Inhibitor Induced Angioedema
Keywords: icatibant; Firazyr; ACE-I
MeSH Terms: interventions — icatibant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icatibant (Experimental): Icatibant at a dose of 30 mg will be administered as a single subcutaneous injection
  Interventions: Drug: Icatibant
- Placebo (Placebo Comparator): Placebo will be administered as a single subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Icatibant — Single dose of 30 mg icatibant administered within 12 hours of the onset of an acute attack of ACE-I-induced angioedema
  Other Names: Firazyr
  Arms: Icatibant
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study is being conducted to compare the safety and efficacy of icatibant with placebo in the treatment for Angiotensin-Converting Enzyme Inhibitor (ACE-I)-Induced Angioedema in Adults.

DETAILED DESCRIPTION:
Angiotensin-converting enzyme inhibitors (ACE-Is) are the class of medications prescribed most frequently for the treatment of hypertension. They are also used post myocardial infarction as well as in patients with heart failure, diabetes mellitus, and chronic kidney disease. Approximately 35 to 40 million patients are on ACE-Is worldwide.

Study HGT-FIR-096 is a multicenter, Phase III, randomized, double-blind, two-armed, placebo-controlled trial. The study population will consist of 118 adult patients, 18 years of age or older, who present with an acute ACE-I-induced angioedema attack. The primary aim of the study is to demonstrate that icatibant is significantly more effective than placebo in resolving attacks of angioedema caused by ACE-I based on the Time to Meeting Discharge Criteria (TMDC). Safety and tolerability, as well as the pharmacokinetics (PK), of icatibant will also be evaluated. Eligible patients will be randomized at a 1:1 ratio to receive a single sub-cutaneous injection of either 30 mg icatibant or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older.
2. Patient is currently being treated with an ACE inhibitor.
3. Patient presenting with an ACE inhibitor-induced angioedema attack of the head and/or neck region within 12 hours of onset (must be sufficiently less than 12 hours to allow study drug to be given with 12 hours of attack onset).
4. Angioedema must be considered at least moderate in severity for at least one of the four angioedema-associated airway symptoms (difficulty breathing, difficulty swallowing, voice changes, tongue swelling).
5. Patient must have voluntarily signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the patient.
6. Females must have a negative urine pregnancy test prior to administration of the study medication, with the exception of those females who have had a total hysterectomy or bilateral oophorectomy, or who are 2 years post-menopausal.

Exclusion Criteria:

1. Patient has a diagnosis of angioedema of other etiology (eg, hereditary or acquired angioedema, allergic angioedema [eg, food, insect bite or sting, evident clinical response to antihistamines and/or corticosteroids], anaphylaxis, trauma, abscess or infection or associated disease, local inflammation, local tumor, post-operative or post-radiogenic edema, salivary gland disorders, other [non-ACE inhibitor] drug-induced angioedema).
2. Patients with a family history of recurrent angioedema.
3. Patients who have had a previous episode(s) of angioedema while not on ACE inhibitor therapy.
4. Patients with acute urticaria (itchy, erythematous wheals).
5. Patients who have an intervention to support the airway (eg, intubation, tracheotomy, cricothyrotomy) due to the current attack of angioedema.
6. Patient has any of the following vascular conditions that, in the judgment of the investigator, would be a contraindication to participation in the study.

   * Unstable angina pectoris or acute myocardial ischemia
   * Hypertensive urgency or emergency (diastolic blood pressure [DBP] >120 mm Hg or systolic blood pressure [SBP] >180 mm Hg)
   * Within 1 month of a stroke or transient ischemic attack
   * New York Heart Association (NYHA) heart failure class IV
7. Patient has a serious or acute condition or illness that, in the judgment of the investigator, would interfere with evaluating the safety and/or efficacy assessments of the study (eg, a condition or illness requiring hemodialysis).
8. Patient is pregnant or breast feeding.
9. Patient has participated in another investigational study in the past 30 days.
10. Patient is unable to understand the nature, scope, and possible consequences of the protocol, or is unlikely or unable to comply with the protocol assessments, or is unlikely to complete the study for any reason.
11. Patients who are not suitable for the study in the opinion of the investigator.
12. Patient has experienced hypersensitivity to the active substance of the investigational product or to any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2015-08-22 (Actual); Study Completion 2015-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (55):
- United States (43):
  - University of California San Diego Medical Center, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Shands Hospital, Gainesville, Florida
  - Orlando Health, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Federal Health Care Center, Chicago, Illinois
  - Cook County Hospital, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Detroit Receiving Hospital and University Health Center, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Inspira Health Network, Vineland, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Weill Medical College of Cornell University, New York, New York
  - East Carolina University, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Hospital - East, Gahanna, Ohio
  - Summit Health, Chambersburg, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - John Peter Smith Hospital, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Ziv Medical Center, Safed
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- United Kingdom (5):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Royal Devon and Exeter Hospital NHS Trust, Exeter
  - University Hospital Aintree, Liverpool
  - Manchester Royal Infirmary, Manchester
  - Queen's Medical Centre, Nottingham

REFERENCES:
- [Result] Sinert R, Levy P, Bernstein JA, Body R, Sivilotti MLA, Moellman J, Schranz J, Baptista J, Kimura A, Nothaft W; CAMEO study group. Randomized Trial of Icatibant for Angiotensin-Converting Enzyme Inhibitor-Induced Upper Airway Angioedema. J Allergy Clin Immunol Pract. 2017 Sep-Oct;5(5):1402-1409.e3. doi: 10.1016/j.jaip.2017.03.003. Epub 2017 May 25. PMID 28552382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 59 sites in the United States, United Kingdom, Israel and Canada.
Pre-assignment Details: Overall 121 participants were randomized, of which 118 received the study medication, and 117 completed the study.
Groups:
- Icatibant 30 mg: Participants received a single dose of icatibant 30 milligram (mg) subcutaneous (SC) injection within 12 hours after the onset of the angiotensin-converting enzyme inhibitor (ACE-I) induced angioedema attack.
- Placebo: Participants received a single dose of placebo matched to icatibant SC injection within 12 hours after the onset of the ACE-I induced angioedema attack.
Period: Overall Study
Arm/Group | Icatibant 30 mg | Placebo
Started | 61 | 60
Completed | 60 | 57
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Icatibant 30 mg: Participants received a single dose of icatibant 30 mg SC injection within 12 hours after the onset of the ACE-I induced angioedema attack.
- Total: Total of all reporting groups
Arm/Group | Icatibant 30 mg | Placebo | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was calculated as the difference between date of birth and date of informed consent, rounded to 1 decimal place.
  years | 60.9 (12.1) | 61.8 (13.4) | 61.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 35 | 62
  Male | 34 | 25 | 59

OUTCOME MEASURES:

1. Primary Outcome: Time to Meeting Discharge Criteria (TMDC)
Description: TMDC was based on the investigator-assessed angioedema-associated upper airway symptom assessments. It was calculated from the time of study drug administration to the earliest time point at which the symptoms of difficulty breathing and difficulty swallowing were absent and the symptoms of voice change and tongue swelling were mild or absent and all subsequent assessments continued to satisfy these conditions. These symptoms were evaluated by the investigator using a 5-point grading scale (0=absent, 1=mild, 2=moderate, 3=severe, and 4=very severe). TMDC was analysed using Kaplan-Meier estimates.
Time Frame: Day 0 up to Day 5
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 61 | 60
days | 4.03 [2.03 to 6.00] | 4.00 [1.03 to 6.00]
Statistical Analysis 1: Comparison: Icatibant 30 mg vs Placebo; A total of 121 participants were analysed, however 3 participants did not receive the study medication and were censored at time 0; Test type: Superiority or Other; p = 0.633, Adjusted Peto-Prentice — Test was performed using a weighted log-rank test called the Peto-Prentice test with a global 2-sided significance level of 5% after adjusting for stratification factors (race, and severity) in the ITT population

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as adverse events/serious adverse events that started or worsened after the study drug treatment.
Time Frame: From start of study drug administration (Day 0) up to follow-up (Day 5)
Population: Safety population included all participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
participants
  Participants with TEAEs | 27 | 21
  Participants with TESAEs | 2 | 1

3. Primary Outcome: Number of Participants With Treatment Emergent Injection Site Reaction
Description: Injection site reaction included erythema, swelling, cutaneous pain, burning sensation, itching and warm sensation
Time Frame: Day 0 to Day 5
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
participants
  Erythema | 31 | 13
  Swelling | 17 | 13
  Cutaneous pain | 10 | 7
  Burning sensation | 15 | 7
  Itching | 13 | 6
  Warm sensation | 16 | 8

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Evaluation, Vital Signs, Electrocardiogram (ECG) and Physical Examination
Description: During laboratory evaluation, serum chemistry and hematology blood tests, and urinalysis were performed. Vital signs parameters included evaluation of pulse rate and systolic and diastolic blood pressure. Standard 12-lead ECGs were performed and ECG recordings were read locally at the study site by a cardiologist. Physical examination was performed with examination of major body systems per routine clinical practice.
Time Frame: Day 0 to Day 5
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
participants | 0 | 0

5. Secondary Outcome: Time to Onset of Symptom Relief (TOSR)
Description: TOSR was calculated for the individual symptoms with pre-treatment scores of 2 (moderate) or more improved by at least 1 severity grade and the individual symptoms with pretreatment scores of 0 or 1 (absent or mild) were scored again at 0 or 1 and all the subsequent assessments continued to satisfy this condition. Time-to-event data were summarized using Kaplan-Meier estimates.
Time Frame: Day 0 up to Day 5
Population: ITT population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 61 | 60
days | 2.00 [0.58 to 3.08] | 1.55 [0.50 to 3.88]

6. Secondary Outcome: Number of Participants Experienced Airway Intervention Due to ACE-I-induced Angioedema
Description: Airway Intervention included intubation, tracheotomy, cricothyrotomy.
Time Frame: Day 0 up to Day 5
Population: Modified Intent to treat (mITT) population included all randomized participants who received the study drug.
Measure: Number; unit: participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
participants | 1 | 0

7. Secondary Outcome: Number of Participants Admitted to Hospital or Intensive Care Unit (ICU)
Description: Number of participants with and without an occurrence of admission to the hospital (inpatient) or ICU post-treatment due to the ACE-I-induced angioedema attack were described.
Time Frame: Day 0 up to Day 5
Population: mITT population.
Measure: Number; unit: participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
participants | 22 | 22

8. Secondary Outcome: Number of Participants Experienced ACE-I-induced Angioedema Attack Following Study Drug Administration
Description: Number of participants with the use of conventional medications (corticosteroids, antihistamines, epinephrine) for the treatment of symptoms of the ACE-I- induced angioedema attack following study drug administration were presented.
Time Frame: Day 0 up to Day 5
Population: mITT population.
Measure: Number; unit: participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
participants | 35 | 35

9. Secondary Outcome: Percentage of Participants With Time to Meeting Discharge Criteria (TMDC) at Specified Time Points
Description: as for outcome 1
Time Frame: 4, 6, and 8 hours post treatment
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Icatibant 30 mg | Placebo
Number analyzed (Participants) | 60 | 58
percentage of participants
  At 4 hours post treatment | 55.0 | 60.3
  At 6 hours post treatment | 78.3 | 75.9
  At 8 hours post treatment | 91.7 | 91.4

10. Other Pre Specified Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Icatibant and Its Metabolites (M1 and M2)
Description: Area under the plasma concentration-time curve of Icatibant and its metabolites (M1 and M2) were analyzed. A population pharmacokinetic analysis approach using sparse pharmacokinetic sampling obtained from a subset of subjects was used to evaluate exposure to icatibant.
Time Frame: 0.75 and 2 hours post-dose
Population: PK analysis population.
Measure: Mean (Standard Deviation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Icatibant 30 mg
Number analyzed (Participants) | 21
hours*nanogram per milliliter (h*ng/mL)
  Icatibant | 2530 (786)
  Metabolite M1 | 2890 (813)
  Metabolite M2 | 3180 (931)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to Day 5
Description: Injection site reactions were reported separately from general reports of adverse events as they were considered as adverse events of special interest.
Arm/Group | Icatibant 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/60 | 1/58
Other Adverse Events (participants affected / at risk) | 14/60 | 11/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icatibant 30 mg (N=60) | Placebo (N=58)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Icatibant 30 mg (N=60) | Placebo (N=58)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 7 (9) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.